CLINICAL TRIAL: NCT04543266
Title: Predicting Metastatic Oral Squamous Cell Carcinomas With Molecular Biomarkers Using Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Choi Siu-wai, Research Assistant Professor, The University of Hong Kong
Other Study IDs: UW19-704
Record Dates: First submitted 2020-09-08; First posted 2020-09-10 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2019-11

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: OSCC; Oral cancer; Machine Learning
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Embedded blocks will be used for protein expressions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Progressive Disease: Patients with metastasis and/or recurrent OSCC were considered as a group of subjects with progressive disease
  Interventions: Procedure: Surgery
- Patients without Progressive Disease: Patients without metastasis and/or recurrent OSCC were considered as a group of subjects without progressive disease
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Resection of tumors
  Other Names: Chemo-radiotherapy

SUMMARY:
Application Management Team:

PI - Siu Wai Choi; email - htswchoi@hku.hk Delegates - Chui Shan Chu; email: sunshine.c@connect.hku.hk FollowUpUsers - Chui Shan Chu; email:sunshine.c@connect.hku.hk

DETAILED DESCRIPTION:
Eligibility Criteria:

- patients were diagnosed with a baseline disease of oral squamous carcinoma.

Exclusion Criteria:

- N/A

Sample size:

- ~500 subjects

Source of Data:

- The data, such as age and medical records, would be obtained from Hospital Authority Clinical Management System (HACMS)

Statistical analysis:

- machine learning will be applied into analysis plan

ELIGIBILITY:
Inclusion Criteria:

* patients with oral squamous carcinoma
* received surgery from 1st October 2000 to 1st October 2019

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective, cohort study of all oral SCC patients who were treated with surgery for their primary oral SCC tumours at Queen Mary Hospital, from 1st October 2000 to 1st October 2019. The investigation will involve retrieval of paraffin embedded tissue blocks, determination of biomarker profile in these tissues, and retrieval of patient data from the Clinical Management System. No new patients will be prospectively recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes of the study are metastasis and recurrent disease | Baseline of OSCC
  These outcomes will be entered as the dependent variables into the machine learning model

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided